CLINICAL TRIAL: NCT07338604
Title: Clinical Study of UTAA07 Injection in the Treatment of CD7 Positive Adult Relapsed/Refractory Hematologic and Lymphatic Systemic Malignancies
Brief Title: Clinical Study of UTAA07 Injection in the Treatment of Hematologic and Lymphatic Systemic Malignancies
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-004-3
Record Dates: First submitted 2025-12-16; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Hematolymphoid Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UTAA07 injection (Experimental)
  Interventions: Drug: CAR-T cell infusion; Drug: UTAA07 injection

INTERVENTIONS:
Drug: CAR-T cell infusion — CAR-T cell infusion
Drug: UTAA07 injection — UTAA07 Injection is a chimeric antigen receptor (CAR)-engineered γδ T-cell product that targets the CD7 antigen expressed on the surface of tumor cells.

SUMMARY:
This is a single-arm, open-label study designed to evaluate the safety, tolerability and cellular pharmacokinetic profiles of UTAA07 Injection. It also aims to preliminarily assess the efficacy of the investigational drug in subjects with relapsed/refractory hematolymphoid malignancies, so as to identify the optimal dose for subsequent formal clinical trials.

DETAILED DESCRIPTION:
This is a single-arm, open-label study designed to investigate the safety, tolerability, and cellular kinetic characteristics of the investigational product. Additionally, it aims to preliminarily observe the efficacy of the investigational product in subjects with relapsed/refractory hematological and lymphoid malignancies, so as to explore the optimal dose for formal clinical applications.

Three dose cohorts are planned, namely 2×10⁹ CAR-γδT cells, 4×10⁹ CAR-γδT cells, and 6×10⁹ CAR-γδT cells. Additional dose cohorts may be added at the discretion of the investigator and/or collaborating institutions. The study will adopt a 3+3 dose escalation/de-escalation schema.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years, regardless of gender.
* Expected survival time ≥ 3 months.
* ECOG performance status score of 0-1.
* Confirmed diagnosis of relapsed/refractory CD7-positive hematolymphoid malignancies at screening.
* Coagulation function, liver and kidney function, and cardiopulmonary function meeting the requirements.
* Ability to understand the trial and signed informed consent form.

Exclusion Criteria:

* A history of malignant tumors other than hematolymphoid malignancies within 5 years prior to screening, excluding carcinoma in situ.
* Positive results for virological tests or syphilis.
* Severe cardiac diseases.
* Unstable systemic diseases as determined by the investigator.
* Active or uncontrolled infections requiring systemic treatment within 7 days prior to screening, excluding mild urinary and reproductive system infections and upper respiratory tract infections.
* Pregnant or lactating women; female subjects planning to become pregnant within 2 years after cell infusion; or male subjects whose partners plan to become pregnant within 2 years after the subject's cell infusion.
* Subjects receiving systemic corticosteroid therapy within 7 days prior to screening, or those judged by the investigator to require long-term systemic corticosteroid therapy during the trial period, excluding inhaled or topical administration.
* Participation in other clinical studies within 1 month prior to screening.
* Evidence of central nervous system (CNS) involvement at screening, such as detection of tumor cells in cerebrospinal fluid (CSF) or imaging findings suggestive of CNS infiltration.
* Patients requiring long-term use of immunosuppressants as determined by the investigator at screening.
* A history of epilepsy or other central nervous system diseases.
* Patients with primary immunodeficiency diseases.
* Other circumstances deemed inappropriate for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 24 months
  Types, frequencies, and severity of adverse events (AEs) and laboratory abnormalities (in accordance with the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] You MJ, Medeiros LJ, Hsi ED. T-lymphoblastic leukemia/lymphoma. Am J Clin Pathol. 2015 Sep;144(3):411-22. doi: 10.1309/AJCPMF03LVSBLHPJ. PMID 26276771